CLINICAL TRIAL: NCT01681576
Title: A Randomized, Double-blind, Crossover Study to Assess the Effects of LCZ696 and Valsartan in Asian Patients With Salt-sensitive Hypertension
Brief Title: Assessment of LCZ696 and Valsartan in Asian Patients With Salt-sensitive Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: CLCZ696A2222
Record Dates: First submitted 2012-08-30; First posted 2012-09-10 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Salt-sensitive Hypertension
Keywords: hypertension, salt sensitivity, valsartan, LCZ696
MeSH Terms: conditions — Hypertension | interventions — Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCZ696 followed by Valsartan (Experimental): Period 1: LCZ696 400mg QD for 4 weeks then washout followed by Period 2: Valsartan 320mg QD for 4 weeks
  Interventions: Drug: Valsartan; Drug: LCZ696
- Valsartan followed by LCZ696 (Experimental): Period 1: Valsartan 320mg QD for 4 weeks then washout followed by Period 2: LCZ696 400mg QD for 4 weeks
  Interventions: Drug: Valsartan; Drug: LCZ696

INTERVENTIONS:
Drug: Valsartan — Valsartan 320mg tablet once daily
Drug: LCZ696 — LCZ696 400mg tablet once daily

SUMMARY:
This study will evaluate the effect of LCZ696 and valsartan on natriuresis, diuresis, and blood pressure in salt-sensitive Asian hypertensive patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent must be obtained before any study assessment is performed.
* Males and females of non-childbearing potential and of legal age (at least 18 years or older as defined by local law).
* Asian patients with mild to moderate essential hypertension, untreated or currently taking antihypertensive therapy with up to two drugs.

Key Exclusion Criteria:

* Women of child-bearing potential.
* History of angioedema, drug-related or otherwise
* History of hypersensitivity to LCZ696, valsartan, or drugs of similar chemical classes.
* Severe hypertension (grade 3 of WHO classification; msDBP ≥100 mmHg and/or msSBP ≥ 180 mmHg) at screening or at the end of the washout period.
* History or evidence of a secondary form of hypertension,
* Transient ischemic cerebral attack (TIA) during the 12 months prior to screening or any history of stroke.
* History of myocardial infarction, coronary bypass surgery or percutaneous coronary intervention (PCI) during 12 month prior to screening.
* Current or history of hypertensive retinopathy.
* Previous or current diagnosis of heart failure (NYHA Class II-IV).
* Clinically significant valvular heart disease at screening.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (3):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Cypress, California
  - Novartis Investigative Site, Glendale, California
- Novartis Investigative Site, Hong Kong, Shatin, NT, Hong Kong
- Novartis Investigative Site, Singapore, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Koyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC

REFERENCES:
- [Derived] Wang TD, Tan RS, Lee HY, Ihm SH, Rhee MY, Tomlinson B, Pal P, Yang F, Hirschhorn E, Prescott MF, Hinder M, Langenickel TH. Effects of Sacubitril/Valsartan (LCZ696) on Natriuresis, Diuresis, Blood Pressures, and NT-proBNP in Salt-Sensitive Hypertension. Hypertension. 2017 Jan;69(1):32-41. doi: 10.1161/HYPERTENSIONAHA.116.08484. Epub 2016 Nov 14. PMID 27849566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1: 4 weeks treatment with LCZ696 400mg QD or Valsartan 320mg, 1-2 weeks wash-out, followed by period 2, 4 weeks treatment with Valsartan 320mg QD or LCZ696 400mg QD
Period: Period 1
Arm/Group | LCZ696 Followed by Valsartan | Valsartan Followed by LCZ696
Started | 36 | 36
Completed | 34 | 36
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Deviation | 1 | 0
Period: Period 2
Arm/Group | LCZ696 Followed by Valsartan | Valsartan Followed by LCZ696
Started | 34 (Period 2: Valsartan 320mg) | 36 (Period 2: LCZ696 400mg)
Completed | 30 | 35
Not Completed | 4 | 1
Not completed — subject/guardian decision | 3 | 1
Not completed — Non-compliance with study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Valsartan 320mg: Period 1: 4 weeks treatment with Valsartan 320mg QD, 1-2 weeks wash-out, followed by period 2, 4 weeks treatment with LCZ696 400mg QD
- Total: Total of all reporting groups
Arm/Group | LCZ696 Followed by Valsartan | Valsartan 320mg | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.5) | 58.9 (7.5) | 57.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Sodium Excretion (Natriuresis) at Day 1
Description: Urine will be collected in fractions of 6 to 24 hours post-dose. From each fraction, a sample will be drawn for analysis of sodium Day 1
Time Frame: 0-6 and 0-24 hours on Day 1
Population: Pharmacodynamic PD analysis set: Patients with any available PD data, who received any study drug and experienced no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: mmol
Groups:
- LCZ696 - ALL: LCZ696 400mg QD
- Valsartan -ALL: Valsartan 320mg QD
Arm/Group | LCZ696 - ALL | Valsartan -ALL
Number analyzed (Participants) | 70 | 67
mmol
  0-6h (n=69,66) | 61.26 (31.167) | 37.13 (20.761)
  0-24h (n=69,66) | 188.87 (74.458) | 138.92 (58.905)

2. Secondary Outcome: Cumulative Sodium Excretion (Natriuresis) at Day 28
Description: Urine will be collected in fractions of 6 to 24 hours post-dose. From each fraction, a sample will be drawn for analysis of sodium Day 28
Time Frame: 0-6 and 0-24 hours on Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol
Groups:
- LCZ696 - ALL: LCZ696 400mg
- Valsartan - ALL: Valsartan 320mg QD
Arm/Group | LCZ696 - ALL | Valsartan - ALL
Number analyzed (Participants) | 70 | 67
mmol
  0-6h (n=69,66) | 39.30 (18.841) | 44.57 (23.479)
  0-24h (n=69,66) | 144.71 (51.094) | 153.82 (62.449)

3. Secondary Outcome: Urine Volume (Diuresis) Over Time
Description: Urine will be collected and volume measured in fractions of 0 to 6 hours and 0 to 24 hours Day-1, Day 1 and Day 28
Time Frame: Day -1, Day 1 & Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | LCZ696 - ALL | Valsartan - ALL
Number analyzed (Participants) | 70 | 67
mL
  Day -1 0-6h (n=70,67) | 855.1 (450.28) | 806.2 (462.20)
  Day -1 0-24h (n=70,67) | 2752.8 (722.53) | 2756.2 (1010.86)
  Day 1 0-6h (n=70,67) | 1215.9 (475.57) | 923.0 (443.65)
  Day 1 0-24h (n=70,67) | 3172.3 (957.70) | 2813.8 (930.05)
  Day 28 0-6h (n=69,66) | 948.8 (415.14) | 1042.7 (530.15)
  Day 28 0-24h (n=69,66) | 2820.0 (847.81) | 3000.2 (1139.75)

4. Secondary Outcome: Seated Office Blood Pressure (BP) (Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)) Over Time
Description: Seated Office BP (systolic blood pressure (SBP) and diastolic blood pressure (DBP))measurements will be performed at trough(immediately prior to dosing at the clinic). Arterial BP readings will be made with an automated BP device.
Time Frame: Day-1, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 - ALL | Valsartan - ALL
Number analyzed (Participants) | 70 | 67
mmHg
  Day -1 Sitting SBP (n=70,67) | 140.20 (13.691) | 137.85 (12.703)
  Day 28 Sitting SBP (n=69,66) | 127.01 (12.723) | 132.07 (15.195)
  Day 14 Sitting DBP (n=69,66) | 80.43 (7.808) | 80.57 (9.246)
  Day 28 Sitting DBP (n=69,66) | 80.44 (7.840) | 81.40 (9.276)
  Day 14 Sitting SBP (n=69,66) | 126.88 (12.451) | 129.23 (12.784)
  Day -1 Sitting DBP (n=70,67) | 86.63 (8.955) | 85.59 (9.299)

5. Secondary Outcome: Mean Sitting Pulse Pressure (PP) Over Time
Description: Sitting mean pulse pressure rate was calculated between ambulatory SBP and DBP measurements
Time Frame: Day-1, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 - ALL | Valsartan - ALL
Number analyzed (Participants) | 70 | 67
mmHg
  Day -1 Sitting mean PP (n=70,67) | 63.91 (8.392) | 64.92 (10.086)
  Day 14 Sitting mean PP (n=69,66) | 71.91 (10.370) | 69.61 (8.888)
  Day 28 Sitting mean PP (n=69,66) | 65.21 (8.999) | 63.63 (8.843)

ADVERSE EVENTS:
Description: Overall, 72 patients with salt-sensitive hypertension were randomized to one of the two crossover treatment arms. For the Safety Set: overall, 71 patients were exposed to at least one dose of LCZ696 400 mg and a total of 67 patients were exposed to at least one dose of valsartan 320 mg.
Groups:
- LCZ696 400 mg QD: LCZ696 400 mg QD
- Valsartan 320 mg QD: Valsartan 320 mg QD
Arm/Group | LCZ696 400 mg QD | Valsartan 320 mg QD
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/67
Other Adverse Events (participants affected / at risk) | 15/71 | 15/67
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 400 mg QD (N=71) | Valsartan 320 mg QD (N=67)
DRY MOUTH (Gastrointestinal disorders) | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 5 | 5
HEADACHE (Nervous system disorders) | 1 | 4
HAEMATURIA (Renal and urinary disorders) | 3 | 2
PYURIA (Renal and urinary disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.